CLINICAL TRIAL: NCT03481894
Title: Prospective, Randomized, Open-Label, Parallel-Group, Active-Controlled, Multicenter Study to Assess Safe and Effective Doses of Kabiven® in Pediatric Patients 2 to 16 Years of Age
Brief Title: Study to Assess Safety and Efficacy of Kabiven® in Pediatric Patients 2 to 16 Years of Age
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: FDA released Fresenius Kabi from this post marketing requirement on 07/16/2019.
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KABI-004-CP3
Record Dates: First submitted 2015-12-03; First posted 2018-03-29 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Malnutrition
Keywords: Parenteral nutrition; Malnutrition; Pediatrics; nutritional needs
MeSH Terms: conditions — Malnutrition; Hyperphagia | interventions — Drugs, Investigational; Drug and Narcotic Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Kabiven® (Experimental): Kabiven is a sterile, hypertonic emulsion in a three chamber container. The separate chambers contain either amino acids with electrolytes, dextrose, or lipid injectable emulsion.
  Interventions: Drug: Kabiven®
- Compounded standard parenteral nutrition (Active Comparator): The control drug will be compounded for each individual patient as prescribed by the physician. Compounding will be performed according to normal hospital procedure which meets the requirements of the United States Pharmacopeial Convention (USP) <797> "Pharmaceutical Compounding-Sterile Preparations".
  Interventions: Drug: Compounded standard parenteral nutrition

INTERVENTIONS:
Drug: Kabiven® — Infusion should start at a low dose (i.e., 12.5 to 25 mL/kg, corresponding to 10.6 to 21.2 kcal/kg/day, 0.49 to 0.98 g lipids/kg/day, 0.41 to 0.83 g amino acids/kg/day and 1.2 to 2.4 g dextrose/kg/day) followed by stepwise increase to the individual target for PN calories.
  The daily dose of the study PN should be infused at a constant rate over 20 to 24 hours.
  Route of Administration: Infusion into a central vein. Duration of Treatment: Study treatment will last for a minimum of 5 and a maximum of 8 consecutive days. Study treatment will be stopped if oral and/or enteral intake covers 80% or more of caloric requirements. If the indication for PN continues after 8 study days, PN will continue per normal institution policy.
  Other Names: Kabiven® for intravenous use (investigational drug)
  Arms: Kabiven®
Drug: Compounded standard parenteral nutrition — Infusion should start at a low dose (i.e., 12.5 to 25 mL/kg, corresponding to 10.6 to 21.2 kcal/kg/day, 0.49 to 0.98 g lipids/kg/day, 0.41 to 0.83 g amino acids/kg/day and 1.2 to 2.4 g dextrose/kg/day) followed by stepwise increase to the individual target for PN calories.
  The daily dose of the study PN should be infused at a constant rate over 20 to 24 hours.
  Route of Administration: Infusion into a central vein. Duration of Treatment: Study treatment will last for a minimum of 5 and a maximum of 8 consecutive days. Study treatment will be stopped if oral and/or enteral intake covers 80% or more of caloric requirements. If the indication for PN continues after 8 study days, PN will continue per normal institution policy.
  Other Names: Compounded standard parenteral nutrition (control drug)
  Arms: Compounded standard parenteral nutrition

SUMMARY:
Demonstrate the safety and efficacy of Kabiven compared to standard parenteral nutrition (PN) administered via central vein in pediatric patients (2 to 16 years of age) requiring PN to meet nutritional needs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 2 to 16 years of age
* Patients who require at least 80% of their caloric intake as PN at study start, and in whom an indication for PN is expected for at least 5 days
* Patients who require a central venous line to receive PN or already have a central venous line in place for other reasons
* Written informed consent from legal representative(s)

Exclusion Criteria:

* Known hypersensitivity to egg, soybean proteins, peanut proteins, corn or corn products, or to any of the active substances or excipients
* Severe hyperlipidemia or severe disorders of lipid metabolism characterized by hypertriglyceridemia (serum triglyceride concentration >1,000 g/dL).
* Inborn errors of amino acid metabolism
* Cardiopulmonary instability (including pulmonary edema, cardiac insufficiency, myocardial infarction, acidosis and hemodynamic instability requiring significant vasopressor support)
* Hemophagocytic syndrome.
* PN in the last 7 days prior to study enrollment.
* Need for chronic PN before study start
* Liver enzymes (either AST, ALT, GGPT), or direct bilirubin exceeding 2 x upper limit of normal range
* Pathologically altered level of any serum electrolyte (sodium, potassium, magnesium, calcium, chloride, phosphate) unless corrected prior to the start of study treatment
* Pathologically altered blood pH, or oxygen saturation, or carbon dioxide unless corrected prior to the start of study treatment
* Pregnancy or lactation
* Participation in another clinical study

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
All adverse events (AE) | After randomization until Day 9
Vital signs: blood pressure | Day 1 - 9
Vital signs: heart rate | Day 1 - 9
Vital signs: body temperature | Day 1 - 9
Vital signs: respiratory rate | Day 1 - 9
Vital signs: saturation of peripheral oxygen (spO2) | Days 1-9
Urine volume | Days 1-9
Change from baseline urea nitrogen on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline alanine aminotransferase (ALT) on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline aspartate aminotransferase (AST) on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline direct bilirubin on days 2, 5 and 9 on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline total bilirubin on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline gamma-glutamyl transpeptidase (GGTP) on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline alkaline phosphatase (ALP) on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline creatinine on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline electrolytes (sodium, potassium, magnesium, calcium, chloride, phosphate) on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline osmolarity on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline pH on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline glucose on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline triglycerides on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline cholesterol on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline lipase on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline amylase on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline total protein on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline c-reactive protein (CRP) on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline white blood cells (WBC) count on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline platelet count on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline red blood cells (RBC) count on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline hemoglobin (hgb) on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline Hematocrit (hct) on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Change from baseline international normalized ratio (INR) on days 2, 5 and 9 | Days 1, 2 (or if not done: Day 3), 5, 9
Nosocomial infection | After randomization until Day 9
  Number of health care associated infections
Need for renal replacement therapy | Days 1-9
Duration of renal replacement therapy | Days 1-9
Need for mechanical ventilation | Days 1-9
Duration of mechanical ventilation | Days 1-9
Change from baseline body weight on days 5 and 9 | Days 1, 5, 9
Change from baseline albumin on days 5 and 9 | Days 1, 5, 9
Change from baseline prealbumin on days 5 and 9 | Days 1, 5, 9
Change from baseline transferrin on days 5 and 9 | Days 1, 5, 9
Change from baseline alpha linolenic acid on days 5 and 9 | Days 1, 5, 9
Change from baseline linoleic acid on days 5 and 9 | Days 1, 5, 9
Change from baseline arachidonic acid on days 5 and 9 | Days 1, 5, 9
Change from baseline eicosatrienoic (mead) acid on days 5 and 9 | Days 1, 5, 9
Change from baseline triene/tetraene ratio (Holman index) on days 5 and 9 | Days 1, 5, 9

CONTACTS AND LOCATIONS:
Overall Officials: Joel D Lim, MD, Principal Investigator — Children's Mercy Hospital, Kansas City, MO 64108
Locations (2):
- United States (2):
  - The University of Chicago Medical Center, Chicago, Illinois
  - Children's Mercy Hospital, Kansas City, Missouri